CLINICAL TRIAL: NCT06042621
Title: Optimizing Time-Limited Trials of Mechanical Ventilation in Acute Respiratory Failure (The TIME Study): A Mixed Methods Observational Study
Brief Title: A Study of Communication Between Clinicians, Patients, and Families in the Intensive Care Unit (ICU)
Acronym: TIME
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2022-1681; 1R01HL168474-01 (NIH); SMPH/MEDICINE/MEDICINE*P (Other: University of Wisconsin-Madison); Protocol Version 10/02/2025 (Other: University of Wisconsin-Madison)
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Respiratory Failure; Mechanical Ventilation; Life-Supporting Treatments; Communication; Decision Making; Critical Care; Palliative Care
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants: Participants will be selected from patients who are admitted to an intensive care unit (ICU) at the University of Wisconsin Hospital, UnityPoint Health - Meriter Hospital, Hospital of the University of Pennsylvania, Penn Presbyterian Medical Center, or Northwestern Memorial Hospital.
- Surrogates: Surrogate participants will be the primary surrogate/s for an eligible patient.
- ICU Team Members: ICU Team Member participants will be members of the hospital staff providing care for an eligible patient.

SUMMARY:
The purpose of this study is to investigate a specific approach to patient care called a time-limited trial (TLT). This approach is sometimes used for people who develop critical illness and are cared for in an intensive care unit (ICU). A time-limited trial is a plan made together by medical teams, patients with critical illness (if they can take part), and their families or other important people helping to make their healthcare decisions. A time-limited trial starts with a discussion of the patient's goals and wishes. Then, a plan is made to use ICU treatments for a set period of time to give the patient the chance to recover. After this time, the patient's response to treatment will be reviewed to help guide what to do next.

Medical teams consider this kind of plan when it is not clear if a patient can recover to a quality of life that is acceptable to them. With a time-limited trial, patients, families, and medical teams experience this uncertainty together.

The main goal of this study is to find the best way to use TLTs for patients in the ICU who have trouble breathing and need mechanical ventilation to help them breathe. The hypothesis is that optimal time-limited trial delivery will reduce the time patients with acute respiratory failure spend in the ICU and will improve the intensive care unit experiences for their families and clinicians.

DETAILED DESCRIPTION:
This is a multi-site observational study that will investigate the time-limited trial approach to care for patients with critical illness, which is a trial of life support with milestones and a timeline to help evaluate whether the patient is improving. The primary objective of this study is to define the optimal care delivery processes of a time-limited trial for adult intensive care unit (ICU) patients who develop acute respiratory failure requiring mechanical ventilation. The two aims of this study are to:

Aim 1: Map the current processes of time-limited trial care delivery for patients with acute respiratory failure.

Aim 2: Elucidate the relationships between time-limited trials, their care delivery processes, and end-of-life outcomes for patients, surrogates, and ICU teams.

For Aim 1, a focused ethnography of approximately 50 time-limited trials will be done to characterize how trials are currently being done in the intensive care unit. This will include direct observation of ICU care provided to patients and real-time interviews with their surrogates and the ICU team members providing their care. Qualitative analyses will be used to characterize TLT activities and team member roles. This data will support the construction of a systems engineering process map, which is a visual tool that diagrams the sequence of process steps and serves as a time-limited trial process measure.

For Aim 2, a prospective cohort of 5,810 patients with acute respiratory failure will be followed to evaluate relationships between time-limited trial exposure and ICU outcomes through a chart review and electronic health record (EHR) data abstraction. The extent to which trial care processes influence surrogate and ICU team member outcomes will be investigated by conducting surveys. Additionally, semi-structured interviews will be conducted with surrogates and ICU team members to investigate how time-limited trial processes work.

The hypothesis is that optimal time-limited trial delivery will reduce intensive care unit length of stay for patients with acute respiratory failure and improve the intensive care unit experiences for their families and clinicians.

ELIGIBILITY:
Inclusion Criteria:

Participants

* Adult (age ≥ 18 years)
* Acute respiratory failure:

  * Hypoxemic (low level of oxygen in the blood) or
  * Hypercapnic (high level of carbon dioxide in the blood)
* Receiving invasive mechanical ventilation (patient needs a breathing machine to help them breathe)

Surrogates

* The main person/s (primary surrogate/s, also known as legally authorized representative/s) who are making medical decisions on behalf of an eligible patient

  * Will be identified by the treating ICU team according to established legal and ethical standards

ICU Team Members

* A member of the interprofessional hospital staff that is caring for an eligible patient

  * Team members may include advanced practice providers (nurse practitioners/ physicians assistants), case managers, chaplains, dietitians, nurses, pharmacists, physical and occupational therapists, physicians (attending/fellow/resident), respiratory therapists, and social workers.

Exclusion Criteria:

Participants

* Participant or their legally authorized representative declines participation or opts-out of data collection

Surrogates

* Cannot complete surveys and interviews in English or Spanish
* Declines participation

ICU Team Members

* Opts out of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from patients who are admitted to an intensive care unit (ICU) at the University of Wisconsin Hospital, UnityPoint Health - Meriter Hospital, Hospital of the University of Pennsylvania, Penn Presbyterian Medical Center, or Northwestern Memorial Hospital. Surrogate participants will be the primary surrogate/s for an eligible patient, and ICU Team Member participants will be members of the hospital staff providing care for an eligible patient.
Sampling Method: Non-Probability Sample
Enrollment: 7818 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Intensive Care Unit (ICU) length of stay | Through participant study completion, an average of 8 days
  Cumulative number of days that participant stays in the intensive care unit.
Surrogate end-of-life intensive care unit (ICU) experience | Between 4 and 16 weeks after participant's hospital discharge
  Surrogate end-of-life intensive care unit (ICU) experience will be measured using the Family Satisfaction in the Intensive Care Unit (FS-ICU) questionnaire. The FS-ICU is a 24 item questionnaire that evaluates family members' satisfaction with their intensive care unit experience. Each question is scored on a 5-point scale from 1 (worst) to 5 (best). The total scores are then converted to a scale from 0 to 100, where 0 is the least satisfied and 100 is the most satisfied.
Intensive Care Unit (ICU) team acute moral distress | Up to 14 days after participant's hospital discharge
  Intensive Care Unit (ICU) team acute moral distress will be measured using the Moral Distress Thermometer (MDT). The MDT first presents a definition of moral distress, then asks the respondent to rate their distress related to a specific context on a 10-point scale from 0 (none) to 10 (worst possible) moral distress.
Direct observation of intensive care unit (ICU) care | Through participant study completion, an average of 8 days
  Direct observations will include observations of interactions that are pertinent to time-limited trials (e.g., daily interprofessional rounds, nursing shift-change handoffs) and family meetings, including both formal (e.g., in a private conference room) or informal (e.g., on medical rounds or at the bedside) discussions between members of the ICU team, surrogates, patients (if able), and other family members. Observations will be documented using field notes, and family meetings will be audio-recorded and transcribed verbatim. Qualitative analysis of field notes and written transcripts will be done to look for themes and trends that emerge from the data.

SECONDARY OUTCOMES:
In-hospital mortality | Through participant study completion, an average of 8 days
  A participant death occurring during the hospital stay.
Length of mechanical ventilation | Through participant study completion, an average of 8 days
  Cumulative number of days that participant receives invasive mechanical ventilation.
Surrogate anxiety and depression | Between 4 and 16 weeks after participant's hospital discharge
  Surrogate anxiety and depression will be measured using the Hospital Anxiety and Depression Scale (HADS), a self-rated scale that aims to measure symptoms of anxiety and depression. The HADS has 14 total items, 7 items measuring anxiety and 7 items measuring depression. Each item is scored on a 4-point Likert scale where scores range from 0 (less anxious or depressed) to 3 (more anxious or depressed).
Patient and family centeredness of care | Between 4 and 16 weeks after participant's hospital discharge
  Patient and family centeredness of care will be measured using the Modified Patient Perceived Patient-Centeredness of Care (PPPC) Scale. The PPPC has 12 total items with a score range of 0 - 100, with higher scores indicating greater patient-centered care.
Surrogate Heard and Understood Measure | Between 4 and 16 weeks after participant's hospital discharge
  The Heard and Understood Measure evaluates the degree to which the surrogate felt heard and understood. This measure has one item with 5 categorical response choices which range from feeling not at all to completely heard and understood by the doctors, nurses and staff in the ICU. Results are summarized by participant counts for each choice.
Surrogate decisional regret | Between 4 and 16 weeks after participant's hospital discharge
  Surrogate decisional regret will be measured using the Decision Regret Scale (DRS) that measures distress or remorse after a health care decision. The DRS has 5 total items scored on a 5-point Likert scale where scores range from 1 (strongly agree) to 4 (strongly disagree). A higher score indicates more regret.
Real-time semi-structured qualitative interviews (Surrogate experience) | Between participant ICU admission and ICU discharge, an average of 8 days
  Serial, real-time interviews will be conducted following an interview guide that will be iteratively revised as necessary during data collection, according to methodological standards of qualitative interview research. The interviews will be audio-recorded and transcribed verbatim.
Semi-structured qualitative interviews (Surrogate experience) | Between 4 and 16 weeks after participant's hospital discharge
  Interviews will be conducted following an interview guide that will be iteratively revised as necessary during data collection, according to methodological standards of qualitative interview research. Surrogate interviews will also use an adapted form of chart-stimulated recall, a case-based interviewing method using prompts to help participants remember and reflect on past events. The interviews will be audio-recorded and transcribed verbatim.
Structured qualitative interviews (ICU team members experience) | Between participant ICU admission and ICU discharge, an average of 8 days
  Brief, real-time structured interviews will collect team members' knowledge, understanding, and approval of time-limited trials for patients in their care.
Semi-structured qualitative interviews (ICU team members experience) | Up to 4 weeks after participant's hospital discharge
  Semi-structured interviews will be conducted following an interview guide that will be iteratively revised as necessary during data collection, according to methodological standards of qualitative interview research. Interviews will also use an adapted form of chart-stimulated recall, a case-based interviewing method using prompts to help participants remember and reflect on past events. The interviews will be audio-recorded and transcribed verbatim.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline M Kruser, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (5):
- United States (5):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - UnityPoint Health - Meriter Hospital, Madison, Wisconsin
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kruser JM, Wiegmann DA, Nadig NR, Secunda KE, Hanlon BM, Moy JX, Ahmad A, Campbell EG, Donnelly HK, Martinez FJ, Polley M, Orhan C, Korth E, Stalter LN, Rowe TJ, Wu AL, Viglianti EM, Eisinger EC, Nguyen O, Halpern SD, Clapp JT. Optimising time-limited trials in acute respiratory failure: a multicentre focused ethnography protocol. BMJ Open. 2025 Dec 14;15(12):e106483. doi: 10.1136/bmjopen-2025-106483. PMID 41397749